CLINICAL TRIAL: NCT06177912
Title: A Phase 3, Randomized, Double-Blind Study to Evaluate the Safety, Tolerability, and Immunogenicity of V116 in Children and Adolescents With Increased Risk of Pneumococcal Disease
Brief Title: A Clinical Study of the V116 Vaccine for Children and Teenagers (V116-013)
Acronym: STRIDE-13
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V116-013; V116-013 (Other: MSD); jRCT2031230559 (Registry Identifier: jRCT); 2023-506236-32 (Registry Identifier: EU CT); U1111-1293-4944 (Registry Identifier: UTN)
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Pneumococcal Infection
MeSH Terms: conditions — Pneumococcal Infections | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- V116 (Experimental): Participants will receive a single 0.5 mL intramuscular (IM) injection of V116 on Day 1
  Interventions: Biological: V116
- PPSV23 (Active Comparator): Participants will receive a single 0.5 mL IM dose of PPSV23 on Day 1.
  Interventions: Biological: PPSV23

INTERVENTIONS:
Biological: V116 — Pneumococcal 21-valent conjugate vaccine with 4 μg of each of the following pneumococcal polysaccharides (PnPs) antigen: 3, 6A, 7F, 8, 9N, 10A, 11A, 12F, 15A, 15C, 16F, 17F, 19A, 20A, 22F, 23A, 23B, 24F, 31, 33F, and 35B in each 0.5 mL sterile solution
  Other Names: Pneumococcal 21-valent Conjugate Vaccine
  Arms: V116
Biological: PPSV23 — Pneumococcal 23-valent conjugate vaccine with 25 μg of each of the following PnPs antigen: 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, and 33F in each 0.5 mL sterile solution
  Other Names: PNEUMOVAX™23
  Arms: PPSV23

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and immunogenicity of V116 compared to PPSV23 in children 2 through 17 years of age. Researchers want to learn if V116 is as good as, or is better than the PPSV23 vaccine in terms of the antibody immune response. V116 and PPSV23 will be studied in children and teenagers who have a higher risk of getting invasive pneumococcal disease (IPD).

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis and stable medical management (for at least 3 months) of one of the following risk conditions for pneumococcal disease: Diabetes mellitus, chronic compensated liver disease, chronic lung disease, chronic heart disease, or chronic kidney disease.
* Has completed pneumococcal conjugate vaccine regimen (PCV7, PCV10, or PCV13) at least 8 weeks before study enrollment.

Exclusion Criteria:

* Has previously received PPSV23 vaccine
* Has a history of active hepatitis within 3 months before study vaccination
* History of invasive pneumococcal disease within 3 years before study vaccination

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 882 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with solicited injection-site adverse events (AEs) | Up to 5 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited injection-site AEs include pain/tenderness, redness/erythema, and swelling.
Percentage of participants with solicited systemic AEs | Up to 5 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited systemic AEs include headache, muscle aches/myalgia, and tiredness/fatigue.
Percentage of participants with vaccine-related serious adverse events (SAEs) | Up to approximately 6 months
  A vaccine-related SAE is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires inpatient hospitalization or prolongs existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is another important medical event.
Geometric Mean Titer of Serotype-specific Opsonophagocytic Activity (OPA) Responses | 30 days postvaccination
  Opsonophagocytic activity (OPA) for the serotypes in V116 will be determined using a multiplexed opsonophagocytic assay (MOPA)

SECONDARY OUTCOMES:
Geometric mean concentrations (GMCs) of serotype-specific Immunoglobulin G (IgG) after vaccination | 30 days postvaccination
  The GMCs for serotype-specific IgG antibodies will be determined using pneumococcal electrochemiluminescence (PnECL)
Geometric mean fold rise (GMFR) from baseline in serotype-specific OPA GMTs | Baseline (Day 1) and Day 30 postvaccination
  The GMFR from baseline in serotype-specific OPA GMTs will be determined using MOPA.
Percentage of participants with ≥4-fold rise from baseline in serotype-specific OPAs GMTs | Baseline (Day 1) and Day 30 postvaccination
  The percentage of participants with ≥4-fold rise from baseline in serotype-specific OPA GMTs will be determined with MOPA.
GMFR from baseline in serotype-specific IgG GMCs | Baseline (Day 1) and Day 30 postvaccination
  The GMFR from baseline in GMCs for serotype-specific IgG antibodies will be determined using PnECL.
Percentage of participants with ≥4-fold rise from baseline in serotype-specific IgG GMCs | Baseline (Day 1) and Day 30 postvaccination
  The percentage of participants with ≥4-fold rise from baseline in serotype-specific IgG GMCs will be determined using PnECL.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (92):
- United States (29):
  - Central Research Associates ( Site 0145), Birmingham, Alabama
  - Velocity Clinical Research, Phoenix ( Site 0122), Phoenix, Arizona
  - Madera Family Medical Group ( Site 0120), Madera, California
  - Optumcare Colorado Springs, LLC ( Site 0113), Colorado Springs, Colorado
  - Accel Research Sites Network- Nona Pediatric Center ( Site 0109), Orlando, Florida
  - University of South Florida-Department of Pediatrics ( Site 0110), Tampa, Florida
  - Velocity Clinical Research at Primary Pediatrics, Macon ( Site 0128), Macon, Georgia
  - Bingham Memorial Hospital ( Site 0149), Blackfoot, Idaho
  - Clinical Research Prime ( Site 0105), Idaho Falls, Idaho
  - Clinical Research Prime Rexburg ( Site 0104), Rexburg, Idaho
  - University of Louisville, Norton Children's Research Institute ( Site 0148), Louisville, Kentucky
  - Velocity Clinical Research, Lafayette ( Site 0103), Lafayette, Louisiana
  - Velocity Clinical Research, Gulfport ( Site 0115), Gulfport, Mississippi
  - Velocity Clinical Research, Hastings ( Site 0114), Hastings, Nebraska
  - Midwest Children's Health Research Institute ( Site 0117), Lincoln, Nebraska
  - Midwest Children's Health Research Institute ( Site 0106), Lincoln, Nebraska
  - Midwest Children's Health Research Institute-Research ( Site 0119), Lincoln, Nebraska
  - Midwest Children's Health Research Institute-Research ( Site 0102), Lincoln, Nebraska
  - Velocity Clinical Research, Albuquerque ( Site 0112), Albuquerque, New Mexico
  - Velocity Clinical Research, Vestal ( Site 0121), Vestal, New York
  - Epic Medical Research - Oklahoma ( Site 0134), Chickasha, Oklahoma
  - Tribe Clinical Research, LLC-Pediatrics ( Site 0118), Greenville, South Carolina
  - Tribe Clinical Research - Spartanburg ( Site 0108), Spartanburg, South Carolina
  - Velocity Clinical Research, Austin ( Site 0129), Austin, Texas
  - PanAmerican Clinical Research ( Site 0132), Brownsville, Texas
  - Epic Medical Research ( Site 0133), DeSoto, Texas
  - Epic Medical Research - Mesquite ( Site 0144), Mesquite, Texas
  - Alliance for Multispecialty Research, LLC ( Site 0140), Layton, Utah
  - Velocity Clinical Research, Salt Lake City ( Site 0124), West Jordan, Utah
- Canada (6):
  - Canadian Center for Vaccinology ( Site 0004), Halifax, Nova Scotia
  - Premier Clinical Trial Network ( Site 0008), Hamilton, Ontario
  - Children's Hospital of Eastern Ontario ( Site 0001), Ottawa, Ontario
  - CHU Sainte-Justine ( Site 0007), Montreal, Quebec
  - McGill University Health Centre - Vaccine Study Centre ( Site 0005), Pierrefonds, Quebec
  - CHU de Québec-Université Laval ( Site 0006), Québec, Quebec
- Chile (5):
  - Centro de Estudios Clínicos (ICIM, Facultad de Medicina Clínica Alemana Universidad del Desarrollo), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile-Pediatric Infectious Diseases and Immunology ( Site 0209), Santiago, Region M. de Santiago
  - Hospital Roberto del Río-Infectología Pediátrica ( Site 0200), Santiago, Region M. de Santiago
  - Hospital Padre Hurtado-NEONATOLOGY/PEDIATRICS ( Site 0204), Santiago, Region M. de Santiago
  - Hospital Dr. Hernán Henríquez Aravena ( Site 0208), Temuco, Región de la Araucanía
- Colombia (4):
  - Clinica Somer ( Site 0405), Rionegro, Antioquia
  - Oncomedica S.A.S ( Site 0402), Montería, Departamento de Córdoba
  - Fundación Valle del Lili ( Site 0404), Cali, Valle del Cauca Department
  - CEIP - Centro de Estudios en Infectología Pediátrica ( Site 0401), Cali, Valle del Cauca Department
- Finland (7):
  - FVR, Kokkolan rokotetutkimusklinikka ( Site 0602), Kokkola, Keski-Pohjanmaa
  - FVR, Oulun rokotetutkimusklinikka ( Site 0600), Oulu, North Ostrobothnia
  - FVR, Tampereen rokotetutkimusklinikka ( Site 0603), Tampere, Pirkanmaa
  - FVR, Seinäjoen rokotetutkimusklinikka ( Site 0604), Seinäjoki, South Ostrobothnia
  - FVR, Turun rokotetutkimusklinikka ( Site 0606), Turku, Southwest Finland
  - FVR, Espoon rokotetutkimusklinikka ( Site 0608), Espoo, Uusimaa
  - MeVac - Meilahti Vaccine Research Center ( Site 0609), Helsinki, Uusimaa
- France (3):
  - Centre Hospitalier Universitaire de Caen - Hôpital Côte de N-Centre de Recherche Clinique Pédiatriq, Caen, Calvados
  - Hôpital Jeanne de Flandre ( Site 0702), Lille, Nord
  - Assistance Publique - Hopitaux de Paris (AP-HP) - Hopital Robert Debre - Centre Hospitalo Universita, Paris
- Israel (3):
  - Rambam Health Care Campus ( Site 0900), Haifa
  - Hadassah Mount Scopus Medical Centre ( Site 0902), Jerusalem
  - Schneider Children's Medical Center ( Site 0903), Petah Tikva
- Japan (8):
  - Saiseikai Yokohamashi Tobu Hospital ( Site 1714), Yokohama, Kanagawa
  - Okinawa Prefectural Nanbu Medical Center and Children's Medical Center ( Site 1701), Kanegusuku, Okinawa
  - Juntendo University Hospital ( Site 1700), Bunkyo-ku, Tokyo
  - Aquakids Clinic ( Site 1709), Edogawa-ku, Tokyo
  - Miyazaki Prefectural Miyazaki Hospital ( Site 1711), Miyazaki
  - University of Miyazaki Hospital ( Site 1705), Miyazaki
  - National Hospital Organization Okayama Medical Center ( Site 1713), Okayama
  - Saitama Prefectural Children's Medical Center ( Site 1702), Saitama
- Poland (5):
  - IN VIVO ( Site 1006), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne Pratia Bydgoszcz ( Site 1004), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckieg-Klinika Pediatrii i Chorob Infekcyjnyc, Wroclaw, Lower Silesian Voivodeship
  - SZPZOZ im. Dzieci Warszawy w Dziekanowie Lesnym ( Site 1007), Łomianki, Masovian Voivodeship
  - Gravita Diagnostyka i Leczenie Niepłodności ( Site 1005), Lodz, Łódź Voivodeship
- Spain (8):
  - Hospital Germans Trias i Pujol ( Site 1104), Badalona, Barcelona
  - Hospital Sant Joan de Déu ( Site 1113), Esplugues de Llobregat, Barcelona
  - Hospital Universitari Vall d'Hebron ( Site 1115), Barcelona, Catalonia
  - CHUS - Hospital Clinico Universitario-Servicio de Pediatría ( Site 1111), Santiago de Compostela, La Coruna
  - Hospital Universitario Severo Ochoa ( Site 1114), Leganés, Madrid
  - Hospital Universitario La Paz-Pediatria y Enfermedades Infecciosas ( Site 1105), Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre-Unidad Pediátrica de Investigación y Ensayos Clínicos ( Site 11, Madrid
  - HOSPITAL UNIVERSITARIO VIRGEN DEL ROCIO ( Site 1112), Seville
- Sweden (3):
  - CTC Karolinska ( Site 1201), Solna, Stockholm County
  - Norrlands universitetssjukhus ( Site 1200), Umeå, Västerbotten County
  - CTC GoCo ( Site 1202), Mölndal, Västra Götaland County
- Thailand (4):
  - Faculty of Medicine Siriraj Hospital-Pediatric Infectious Diseases ( Site 1601), Bangkoknoi, Bangkok
  - Chulalongkorn University-Pediatrics ( Site 1602), Pathumwan, Bangkok
  - Faculty of Tropical Medicine, Mahidol University - Vaccine Trial Centre ( Site 1604), Ratchathewi, Bangkok
  - Songklanagarind hospital-Department of Pediatrics ( Site 1603), Hat Yai, Changwat Songkhla
- Turkey (Türkiye) (7):
  - Çukurova Üniversitesi Tıp Fakültesi Adana Hastanesi-Pediatric Infection ( Site 1302), Sarçam, Adana
  - Hacettepe Universite Hastaneleri ( Site 1300), Ankara
  - Ankara Universitesi Tip Fakultesi Hastanesi ( Site 1304), Ankara
  - Ankara Bilkent Şehir Hastanesi-Infectious Disease and Clinical Microbiology ( Site 1301), Ankara
  - Sisli Etfal Training and Research Hospital ( Site 1305), Istanbul
  - Ege Universitesi Hastanesi ( Site 1306), Izmir
  - Erciyes Universitesi Tıp Fakultesi Hastaneleri-pediatric infection ( Site 1303), Kayseri

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26202&tenant=MT_MSD_9011